CLINICAL TRIAL: NCT00523796
Title: InPractice Survey on the Treatment of Hypercholesterolemia
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Other Study IDs: NIS-CVN-CRE-2007/1; VN-NIS-0001 (Other: NIS Registry)
Record Dates: First submitted 2007-08-30; First posted 2007-09-03 (Estimated); Last update posted 2011-02-16 (Estimated); Status verified 2011-02

CONDITIONS: Hypercholesterolemia
Keywords: dyslipidemia; in practice survey; Vietnam
MeSH Terms: conditions — Hypercholesterolemia; Dyslipidemias

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a multi-centre survey of patients who are currently on lipid-lowering pharmacological treatment. Data collection for each patient will take place at one visit.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 years of age or older of either sex.
* Subject is on lipid-lowering drug treatment for at least 3 months, with no dose change for a minimum of 6 weeks.

Exclusion Criteria:

* Subjects who are unwilling or unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2007-02; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pham Gia Khai, Prof, Study Chair — Vietnamese Cardiovascular Association; Nguyen Manh Phan, Prof, Study Chair — Vietnamese Cardiovascular Association; Than Trong Son, MD, Study Director — AstraZeneca
Locations (1):
- Research Site, Hanoi, Vietnam